CLINICAL TRIAL: NCT03311854
Title: A Pilot, Open-label, Single Arm, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous Administrations of Emapalumab, an Anti-interferon Gamma (Anti-IFNγ) Monoclonal Antibody, in Patients With Systemic Juvenile Idiopathic Arthritis (sJIA) or Adult-onset Still's Disease (AOSD) Developing Macrophage Activation Syndrome/Secondary HLH (MAS/sHLH)
Brief Title: A Study to Investigate the Safety and Efficacy of Emapalumab, an Anti-IFN-gamma mAb in Patients With Systemic Juvenile Idiopathic Arthritis (sJIA) or Adult-onset Still's Disease (AOSD) Developing Macrophage Activation Syndrome/Secondary HLH (MAS/sHLH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0501-06
Record Dates: First submitted 2017-08-21; First posted 2017-10-17 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Macrophage Activation Syndrome; Lymphohistiocytosis, Hemophagocytic; Arthritis, Juvenile; Adult Onset Still Disease
Keywords: Emapalumab; Gamifant; Macrophage activation syndrome; Secondary hemophagocytic lymphohistiocytosis; Interferon-gamma; Systemic juvenile idiopathic arthritis; Adult-onset Still's disease; MAS; HLH; sHLH; IFN-gamma; IFNγ; sJIA; AOSD; NI-0501-06; NI-0501
MeSH Terms: conditions — Macrophage Activation Syndrome; Lymphohistiocytosis, Hemophagocytic; Arthritis, Juvenile; Still's Disease, Adult-Onset | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental)
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Emapalumab was administered at an initial dose of 6 mg/kg by intravenous infusion. Emapalumab treatment continued at a dose of 3 mg/kg, every 3 days until study day 15, and then twice-a-week for an additional 2 weeks, i.e., until study day 28. The emapalumab regimen could be adapted (the frequency between infusions shortened, the dose increased, or the treatment prolonged beyond 4 weeks) upon assessment of a favourable benefit-risk profile. There was a 4-week off-drug follow-up period (up to Week 8).
  Other Names: Gamifant

SUMMARY:
Macrophage Activation Syndrome (MAS) is a rare, life-threatening condition characterized by uncontrolled hyperinflammation which may develop on the background of systemic Juvenile Idiopathic Arthritis (sJIA) or Adult-onset Still's Disease (AOSD). Emapalumab is a monoclonal antibody neutralizing interferon-gamma (IFN-gamma), a key cytokine which contributes to the inflammation and tissue damage seen in MAS. The purpose of this study is to assess the safety, tolerability and efficacy of emapalumab in sJIA or AOSD participants developing MAS, presenting an inadequate response to high dose glucocorticoid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* For sJIA patients: Confirmed sJIA diagnosis. For patients presenting with MAS in the context of the onset of sJIA, high presumption of sJIA will suffice for eligibility. For AOSD patients: confirmed AOSD diagnosis as per Yamaguchi criteria.
* Diagnosis of active MAS.
* An inadequate response to high dose i.v. glucocorticoid treatment administered for at least 3 days as per local standard of care (including but not limited to pulses of 30 mg/kg PDN on 3 consecutive days). High dose i.v. glucocorticoid should not be lower than 2 mg/kg/day of PDN equivalent in 2 divided doses (or at least 60 mg/day in patients of 30 kg or more). In case of rapid worsening of the patient's condition and/or lab parameters, inclusion may occur within less than 3 days from starting high dose i.v. glucocorticoids.
* Tocilizumab, TNF inhibitors and canakinumab, if administered, have to be discontinued before emapalumab initiation.
* Having received guidance on contraception for both male and female patients sexually active and having reached puberty. Females of child-bearing potential require use of highly effective contraceptive measures. Males with partners(s) of child-bearing potential must agree to take appropriate precautions.
* Informed consent provided by the patient (as required by local law), or by the patient's legally authorized representative(s) with the assent of patients who are legally capable of providing it, as applicable.

Exclusion Criteria:

* Diagnosis of suspected or confirmed primary HLH or HLH consequent to a neoplastic disease.
* Active mycobacteria (typical and atypical), Histoplasma Capsulatum, Shigella, Salmonella, Campylobacter and Leishmania infections.
* Clinical suspicion of latent tuberculosis.
* Positive serology for HIV antibodies.
* Presence of malignancy.
* Patients who have another concomitant disease or malformation severely affecting the cardiovascular, pulmonary, CNS, liver or renal function that in the opinion of the Investigator may significantly affect likelihood to respond to treatment and/or assessment of emapalumab safety.
* History of hypersensitivity or allergy to any component of the study drug
* Receipt of a BCG vaccine within 12 weeks prior to screening.
* Receipt of live or attenuated live vaccines (other than BCG) within 6 weeks prior to screening.
* Pregnant or lactating female patients.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Cincinnati Children'S Hospital, Cincinnati, Ohio, United States
- Hôpital Necker-Enfants Malades, Unité d'Immunologie-hématologie et Rhumatologie pédiatriques, Paris, France
- IRCCS Ospedale Pediatrico, Bambino Gesù, Rome, Italy
- Hospital Sant Joan de Deu, Barcelona, Spain
- Great Ormond Street Hospital for Children, London, United Kingdom

REFERENCES:
- [Derived] Brossard P, Laveille C. Population Pharmacokinetics of the Anti-Interferon-Gamma Monoclonal Antibody Emapalumab: An Updated Analysis. Rheumatol Ther. 2024 Jun;11(3):869-880. doi: 10.1007/s40744-024-00669-y. Epub 2024 Apr 25. PMID 38662147
- [Derived] De Benedetti F, Grom AA, Brogan PA, Bracaglia C, Pardeo M, Marucci G, Eleftheriou D, Papadopoulou C, Schulert GS, Quartier P, Anton J, Laveille C, Frederiksen R, Asnaghi V, Ballabio M, Jacqmin P, de Min C. Efficacy and safety of emapalumab in macrophage activation syndrome. Ann Rheum Dis. 2023 Jun;82(6):857-865. doi: 10.1136/ard-2022-223739. Epub 2023 Mar 31. PMID 37001971

RESULTS

PARTICIPANT FLOW:
Groups:
- All Treated Population: Of the 16 patients who were screened for the study, 14 were enrolled. All 14 patients completed the study; no patient was withdrawn after the start of treatment. All 14 patients received emapalumab and were included in the all treated population.
Period: Overall Study
Arm/Group | All Treated Population
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: Baseline data are provided for all participants who were enrolled in the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
  Italy | 7
  United Kingdom | 2
  Spain | 1
  France | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence, Severity, Causality, and Outcomes of AEs (Serious and Nonserious)
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Groups:
- All Treated Population: The all treated population included all patients who received any part of an infusion of emapalumab.
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants
  Number of participants with a TEAE | 13
  Number of participants with a serious TEAE | 6
  Number of participants with a severe TEAE | 2
  Number of participants with a moderate TEAE | 10
  Number of participants with a mild TEAE | 13
  Number of participants with a TEAE related to emapalumab | 4
  Number of participants with a TEAE unrelated to emapalumab | 13
  Number of participants with a TEAE with an outcome of recovered/resolved | 13
  Number of participants with a TEAE with an outcome of not recovered/not resolved | 3
  Number of participants with a TEAE with an outcome of recovering/resolving | 1
  Number of participants with a TEAE with an outcome of unknown | 1

2. Primary Outcome: Evolution of Laboratory Parameters
Description: Shifts from baseline in the following MAS-relevant laboratory parameters are reported:
  * Leukocytes
  * Platelets
  * Lactate dehydrogenase (LDH)
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Ferritin
  * C-reactive protein
  * Activated partial thromboplastin time (aPTT)
  * Prothrombin time
  * D-dimer
  * Fibrinogen
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants
  Leukocytes: From a high value at baseline to a value within the reference range at Week 8 | 2
  Leukocytes: From a low value at baseline to a value within the reference range at Week 8 | 4
  Leukocytes: From a low value at baseline to a high value at Week 8 | 2
  Platelets: From a high value at baseline to a value within the reference range at Week 8 | 1
  Platelets: From a low value at baseline to a value within the reference range at Week 8 | 6
  Platelets: From a low value at baseline to a high value at Week 8 | 3
  LDH: From a high value at baseline to a value within the reference range at Week 8 | 6
  ALT: From a high value at baseline to a value within the reference range at Week 8 | 10
  ALT: From a high value at baseline to a low value at Week 8 | 1
  AST: From a high value at baseline to a value within the reference range at Week 8 | 11
  Ferritin: From a high value at baseline to a value within the reference range at Week 8 | 11
  Ferritin: From a high value at baseline to a low value at Week 8 | 2
  C-reactive protein: From a high value at baseline to a value within the reference range at Week 8 | 9
  aPTT: From a high value at baseline to a value within the reference range at Week 8 | 1
  aPTT: From a high value at baseline to a low value at Week 8 | 1
  aPTT: From a value within the reference range at baseline to a low value at Week 8 | 3
  aPTT: From a low value at baseline to a value within the reference range at Week 8 | 1
  aPTT: From a low value at baseline to a high value at Week 8 | 1
  Prothrombin time: From a high value at baseline to a value within the reference range at Week 8 | 5
  Prothrombin time: From a high value at baseline to a low value at Week 8 | 1
  Prothrombin time: From a value within the reference range at baseline to a low value at Week 8 | 3
  Prothrombin time: From a low value at baseline to a value within the reference range at Week 8 | 1
  D-dimer: From a high value at baseline to a value within the reference range at Week 8 | 8
  Fibrinogen: From a high value at baseline to a value within the reference range at Week 8 | 1
  Fibrinogen: From a value within the reference range at baseline to a high value at Week 8 | 1
  Fibrinogen: From a low value at baseline to a value within the reference range at Week 8 | 5
  Fibrinogen: From a low value at baseline to a high value at Week 8 | 1

3. Primary Outcome: Number of Participants Withdrawn Due to Safety Reasons
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 0

4. Primary Outcome: Number of Participants Achieving MAS Remission at Week 8 After Initiation of Emapalumab Treatment
Description: Remission from MAS was evaluated according to the following criteria:
  Resolution of clinical signs and symptoms according to the investigator (MAS clinical signs and symptoms activity score ≤ 1)
  and
  Normalization of laboratory parameters relevant to MAS, as follows:
  * WBC count and platelet count above the LLN.
  * LDH below 1.5 × the ULN.
  * ALT and AST both below 1.5 × the ULN.
  * Fibrinogen higher than 100 mg/dL.
  * Ferritin levels decreased by at least 80 % from values at screening or baseline (whichever was higher) or below 2000 ng/mL, whichever was lower.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 11

5. Primary Outcome: Time to First MAS Remission
Time Frame: Up to Week 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
days | 25 [19 to 56]

6. Primary Outcome: Number of Participants for Whom Glucocorticoids Could be Permanently Tapered at Any Time During the Study
Description: Permanently tapering by at least 50% of the equivalent dose of prednisone. This was defined as achieving reduction of 50% of the baseline dose [SD0] and maintaining the reduction until the end of study).
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 12

7. Primary Outcome: Time to Achievement of Permanent Glucocorticoids Tapering
Description: Time to achievement of permanent glucocorticoid tapering by at least 50% of the equivalent dose of prednisone administered at emapalumab treatment start.
Time Frame: Up to Week 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
days | 14.5 [4 to 28]

8. Primary Outcome: Survival Time
Description: Number of participants alive at the end of the study
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 14

9. Primary Outcome: Number of Participants Withdrawn From the Study Due to Lack of Efficacy
Description: Number of participants withdrawn from the study due to lack of efficacy
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 0

10. Primary Outcome: Levels of Emapalumab Concentration
Description: On all infusion days, PK samples were collected before the infusion start and between 15 and 30 minutes after infusion completion. In addition, following the first emapalumab infusion, PK samples were collected approximately 24 and 48 hours post-infusion, and following the second emapalumab infusion, PK samples were collected approximately 48 hours post-infusion. Upon treatment completion, PK samples were collected on all non-infusion visits until the 4-week follow-up visit/EOS.
Time Frame: Data from the following time points are presented: SD0 (pre- and post-dose), Week 4 Visit 2 (pre- and post-dose), and 4-week follow-up visit/EoS.
Population: Emapalumab concentrations were below the detection limit for all patients at SD0, except for Patient 501-001, in whom the emapalumab concentration (pre-dose) was 62108.4 μg/L. It should be noted that on SD1, the measurement results of emapalumab were below the detection limit for Patient 501-001, so it could not be ruled out that the samples from SD0 and SD1 for this patient were interchanged.
Measure: Mean (Standard Deviation); unit: μg/L
Groups:
- All Treated Population: The all treated population included all patients who received any part of an infusion of emapalumab.
  Note: the Week 4 Visit 2 (post-dose) emapalumab concentration levels were based on 7 participants.
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
μg/L
  Study Day 0 (pre-dose) | 5455.444 (19985.0660)
  Study Day 0 (post-dose) | 104740.254 (20994.1054)
  Week 4 Visit 2 (pre-dose) | 115472.076 (58676.7953)
  Week 4 Visit 2 (post-dose) | 212900.657 (87466.3031)
  4-week follow-up Visit/EoS | 46447.462 (33657.0174)

11. Primary Outcome: Pharmacodynamic Parameters
Description: Levels of total INF-gamma, CXCL9 and CXCL10
Time Frame: Up to Week 8
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- All Treated Population: Study Day 0: Levels measured pre-dose on Study Day 0 in participants in the all treated population which included all patients who received any part of an infusion of emapalumab.
- All Treated Population: 4-week Follow-up Visit/EoS: Levels measured at the 4-week follow-up visit/EoS in participants in the all treated population which included all patients who received any part of an infusion of emapalumab.
Arm/Group | All Treated Population: Study Day 0 | All Treated Population: 4-week Follow-up Visit/EoS
Number analyzed (Participants) | 14 | 14
ng/L
  CXCL9 | 21986.010 (29405.8787) | 255.654 (596.4149)
  CXCL10 | 7935.418 (9115.2857) | 639.102 (1058.9589)
  Total IFN-γ | 425.528 (1191.8391) | 2132.656 (2967.4920)

12. Primary Outcome: Number of Participants Who Demonstrated a Presence of Circulating Antibodies Against Emapalumab to Determine Immunogenicity
Description: The presence of circulating antibodies against emapalumab was inferred by positive results for anti-drug antibodies (ADAs).
Time Frame: Up to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated Population
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded in patients from Study Day 0 (the day of the first emapalumab administration), during emapalumab treatment, and up to and including the 4-week follow-up visit/end of study (a minimum duration of 56 days). All adverse events were followed up for outcome at end of study; all serious adverse events were followed up until resolution.
Description: While all adverse events reported by the participants or their relatives or observed by the Investigator or their staff during the clinical study from the signature of the informed consent form up to and including the end-of-study visit were recorded, only treatment-emergent adverse events (those that occurred after the start of the first emapalumab administration) are reported here.
Arm/Group | All Treated Population
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Population (N=14)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Juvenile myoclonic epilepsy (Nervous system disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Still's disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Population (N=14)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 3 (3)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (4)
Axonal neuropathy (Nervous system disorders) | 1 (1)
Juvenile myoclonic epilepsy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Catheter site thrombosis (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (4)
Secretion discharge (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Eye oedema (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Adenovirus test positive (Investigations) | 1 (1)
BK polyomavirus test positive (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1)
Respirovirus test positive (Investigations) | 1 (1)
Still's disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT03311854/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT03311854/SAP_001.pdf